CLINICAL TRIAL: NCT04004117
Title: Effect of Sublingual Fentanyl on Breathlessness in COPD : A Randomized Cross-over Trial
Brief Title: Effect of Sublingual Fentanyl on Breathlessness in COPD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jean Bourbeau, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIMUHCCOPDJB
Record Dates: First submitted 2019-05-27; First posted 2019-07-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Multicentered randomized clinical trial, triple-blinded, cross-over design, comparing fentanyl sublingual at a dose 12,5 mcg to placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All research staff, treating clinicians, analysts and patients will remain blinded to the treatment allocation.
  Unbinding will only occur in emergency situations following consultation with the principal investigator and at the conclusion of collecting the last data point for the last participant in the entire study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl s/l (Experimental): Sublingual fentanyl will consist in liquid fentanyl at a concentration of 25 mcg/mL, with preparation by the pharmacist of pre-dosed syringes of 12,5 mcg (0,5 mL).
  Interventions: Drug: Fentanyl citrate solution sublingual; Drug: Placebo oral liquid
- Placebo (Placebo Comparator): Placebo will consist in simple syrup (simple syrup B.P. - NPN: 00050121) administered sublingually with syringe.
  Interventions: Drug: Fentanyl citrate solution sublingual; Drug: Placebo oral liquid

INTERVENTIONS:
Drug: Fentanyl citrate solution sublingual — Solution of fentanyl citrate (DIN : 02384124 / 02240434 / 02385406) will be administered sublingually by syringe. The dose is 12,5 mcg.
Drug: Placebo oral liquid — Placebo will consist in simple syrup (simple syrup B.P. - NPN: 00050121) administered sublingually with syringe.

SUMMARY:
There is actually no physiologic or clinical data in the literature to clearly define the potential benefits and side effects of sublingual fentanyl in patients with COPD. Therefore, the purpose of this study is to test the hypothesis that sublingual fentanyl will improve exercise capacity and dyspnea control in severe COPD patients experiencing persistent breathlessness despite optimal management.

DETAILED DESCRIPTION:
The purpose of this study is to test the hypothesis that sublingual fentanyl will improve exercise capacity and dyspnea control in severe COPD patients experiencing persistent breathlessness despite optimal management.

To demonstrate the effectiveness of sublingual fentanyl, the investigators suggest a dose of 12,5 mcg. The investigators base this decision on several considerations :

* Local practice and experience : the safety of a dose of 12,5 mcg of sublingual fentanyl has been show in the investigators local experience (see section 1.3 Clinical experience with fentanyl).
* Although there is not enough information to determine the exact equivalence between sublingual fentanyl and oral morphine, the conversion between intravenous fentanyl and oral morphine can be done. Based on the monograph of fentanyl citrate, 10 mcg of intravenous fentanyl citrate are equivalent to 10 mg of intravenous morphine, which are equivalent to 20 to 30 mg of oral morphine. Subsequently, 12,5 mcg of sublingual fentanyl may be equivalent to a oral morphine dose between 2,5 and 3,75 milligrams. This represent a smaller dose than the dose of 0,1 mg/kg oral morphine that was demonstrated to be safe in a recent study done by a group at McGill in a severe COPD population (Abdallah et al. Eur Respir J 2017; 50: 1701235).
* The study will only include patients who are already on morphine, because they represent the target population and have less risk of adverse events than an opioid-naive population.
* To ensure safety, participants will be actively monitored during the study. A doctor will be present at administration of the drug and the antidote, naloxone, will be readily available if needed. Participants will be monitored on-site for 30 minutes after completion of CPET and discharge only if no evidence of side effects. Participants will be informed to not drive for 24 hours following each period of treatment. A phone call follow-up will be done 24-48 hours after treatment visits.

General Objective:

The general objective is to demonstrate the role of sublingual fentanyl liquid to improve exertional shortness of breath in patients with severe to very severe COPD.

Primary Objective :

The primary objective is to evaluate in severe/very-severe COPD the effect of 12,5 mcg fentanyl sublingual liquid as compared with placebo, on i) post-dose difference in exertional breathlessness at isotime (Isotime definition : highest equivalent 2 min interval of exercise completed by a given participant) ii) Post-dose difference in exercise endurance time (EET)

The study is a multicentred randomized clinical trial, triple-blinded, cross-over design, comparing fentanyl sublingual at a dose 12,5 mcg to placebo in severe/very-severe COPD already taking low dose of morphine because of refractory dyspnea.

To detect a minimally clinically important (MCID) difference of 1 Borg unit (40) at iso-time between treatments, we assume an α of 0.05 and a within-subject standard deviation of 1 Borg unit: a total of 20 patients will provide >80% power; assuming an attrition rate of 20%, a total of 24 patients will be recruited for this study.

All data will be de-nominalized in order to respect privacy. Data will be collected in an anonymous data sheet, protected by a password. Only investigators and statistician will have access to this data sheet.

The principal analysis of the relative change in dyspnea intensity at iso-time (primary end-point) after treatment with morphine sulfate vs. placebo will be conducted using an unadjusted paired t-test. Secondary analyses to assess treatment responses on secondary end-points (e.g. arterialized capillary PCO2, EET, dyspnea unpleasantness, ventilation, breathing pattern, operating lung volumes, etc.) will be done using paired t-tests adjusted (Bonferroni) for multiple comparisons. Pearson correlations will be used to establish associations between intra-subject post-dose differences in iso-time dyspnea intensity ratings and relevant independent variables (e.g. arterialized capillary PCO2, ventilation, breathing pattern, MDP results, etc.) and various baseline patient characteristics (possible covariates). Stepwise multiple regression analysis will then be carried out with significant independent variables and relevant covariates.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 40 years
* Cigarette smoking history ≥10 pack years
* Clinical diagnosis of severe to very severe COPD, i.e. post-β2-agonist FEV1 <50% and FEV1/FVC <0.70
* Chronic activity-related dyspnea, define as any one or combination of a modified MRC of 3-4 or a BDI focal score ≤ 8
* Uncontrolled daily activity-related dyspnea despite optimal medical treatment, including oral morphine treatment at a dose of a least 4 mg per day
* No change in medication dosage or frequency of administration in the previous 2 weeks
* No exacerbations or hospitalizations in the preceding 4 weeks

Exclusion Criteria:

* CO2 retention, defined as a resting arterial/capillary PCO2 of >50 mmHg
* Self-reported history of addiction/substance abuse
* Acute alcoholism
* Presence of important contraindications to cardiopulmonary exercise testing (CPET)
* History of hypersensitivity to fentanyl or any component of the formulation
* Actual use of methadone
* Concurrent use or use within 14 days of a monoamine oxidase (MAO) inhibitor
* Severe CNS depression
* Convulsive disorders
* Known or suspected mechanical GI obstruction (e.g., bowel obstruction or strictures) or any diseases/conditions that affect bowel transit (e.g., ileus of any type)
* Increased cerebrospinal or intracranial pressure and head injury
* Active mouth mucositis
* Dementia diagnosis or significant neurocognitive problems
* History of severe chronic kidney disease (stage 4-5)
* Women of child bearing potential (defined as not having gone at least 12 months without a menstrual period) will be required to take a routine (urine) pregnancy test to rule out the possibility of pregnancy
* Breast-Feeding women
* Acute or unstable, clinically significant abnormal findings in physical exam, vital signs or ECG (as per Investigators opinion)
* Patients receiving long-term treatment with Oxygen >4.0 liters/minute (L/min). They must be ambulatory and be able to attend clinic visits. While breathing supplemental oxygen, they must demonstrate an oxyhemoglobin saturation ≥ 89%.
* Malignancy, current or within the past 2 years. that the patient is not stable
* Scheduled major surgical procedure during the course of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Breathlessness | Up to 10 days after visit 1
  Post-dose difference in exertional breathlessness at isotime (isotime definition : highest equivalent 2 min interval of exercise completed by a given participant).
Exercise capacity | Up to 10 days after visit 1
  Post-dose difference in exercise endurance time (EET)

SECONDARY OUTCOMES:
Number and description of adverse effects | Up to 48 hours after treatment administration
  Number and description of adverse effects
Locus of Symptoms | Up to 10 days after visit 1
  Percentage contribution of breathlessness and leg discomfort to exercise cessation
Qualitative descriptors of breathlessness at end exercise | Up to 10 days after visit 1
  Description by patients of the characteristics of breathlessness at the end of exercise
Change in multidimensional evaluation of dyspnea | Up to 10 days after visit 1
  Evaluation of the multidimensional components of dyspnea following each intervention and using the Multidimensional Dyspnea Profile (MDP) questionnaire. The questionnaire contains a total of 11 questions to characterize dyspnea. Each questions is a symptom or a sensation that need to be rated on scale from 0 to 10 depending on the intensity of the symptom/sensation, with 0 representing the absence of symptom and 10 representing the higher perception of symptom. There is no combination to form a total score.
Participant blinded preference | Up to 10 days after visit 1
  At the last visit, the investigators will ask to patients which intervention they preferred regarding relief of breathlessness and comfort during exercise
Difference in the locus of symptoms limiting exercise during a cardio-pulmonary exercise test response when comparing responders to non-responders. | Up to 10 days after visit 1
  Responders will be define as participant with ≥ 1-point improvement in Borg dyspnea. The locus of symptom is the symptom that limit the exercise test (breathlessness, leg fatigue or both).

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bourbeau, MD, Principal Investigator — Reseach Institute MUHC
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to have the data share by other researcher. All data will be denominalized in order to respect privacy. Data will be collected in an anonymous data sheet, protected by a password. Only investigators and statistician will have access to this data sheet.